CLINICAL TRIAL: NCT06774521
Title: Effectiveness of Pilates Exercises in the Treatment of Dysmenorrhea: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Doç.Dr.Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar19
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Methionine Adenosyltransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): those who did not receive any intervention
  Interventions: Other: control
- reformer exercise group (Experimental): They will practice reformer pilates exercises
  Interventions: Other: reformer
- mat exercise group (Experimental): They will practice mat pilates exercises
  Interventions: Other: mat

INTERVENTIONS:
Other: control — There is no intervention
  Arms: control group
Other: reformer — Reformer exercises:
  Foodwork Swan Short Spin Long Stretch Keen Stretch Hug Tree Bridge Pulling Straps Short Box Abdominal Hundred Twist Star
  Arms: reformer exercise group
Other: mat — Mat exercises:
  Neck exercises Trunk stabilization exercises Shoulder exercises Posture exercises
  Arms: mat exercise group

SUMMARY:
The aim of this study is to investigate the effectiveness of Pilates exercises in the treatment of dysmenorrhea and to contribute to the literature and information on this subject.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. The study will be conducted at the Fizyorapt physiotherapy and exercise consultancy center. It will be divided into 2 main groups as those between the ages of 18-50, those with a menstrual period of 3-9 days, those with menstrual pain complaints, and those who cooperate in completing the assessment scales. Participants will be asked to continue the given exercises for 6 weeks, 2 days a week and 45 minutes. People with psychological and physical disabilities will not be included in regular exercise. A personal information form will be prepared by the researcher in order to collect data on the sociodemographic characteristics of the participants. Visual analog scale (VAS) will be used to measure pain intensity and pain relief, Beck depression scale to determine depression symptoms, and menstruation symptom scale to evaluate menstrual pain and symptoms. These surveys will be repeated before and at the end of the study. The data to be obtained will be evaluated using the SPSS24 package program.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals between the ages of 18-50
* Those with a menstrual period of 3-9 days
* Having menstrual pain complaints in most of their menstrual cycles
* Cooperating in completing the assessment scales

Exclusion Criteria:

* Having a history of abdominal surgery
* Having an active infection
* Having knee pain

  -. Using medication
* Participants with any pathology that prevents exercise will not be included in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 14 weeks
  Participants were included in the "healthy" category when they marked the 0-1 range of the scale, and were included in the "Menstruation pain" category when they marked the 1.1-10 range. They were divided into 3 groups according to pain severity. 1.1-3: Mild pain, 3.1-7: Moderate pain, 7.1-10: Severe pain.
Menstruation Symptom Scale | 14 weeks
  It is a 5-point Likert-type scale and consists of three sub-parameters: 'negative effects/somatic effects', 'menstrual pain' and 'coping methods', and 22 items. The person is asked to give a score between '1' never and '5' always for the symptoms they experience related to menstruation. The Menstruation Symptom Scale (MSS) score is calculated by taking the total score average. An increase in the mean score indicates an increase in the severity of menstrual symptoms.
Fatigue Severity Scale | 14 weeks
  It consists of 9 questions. Each question is scored between 1 and 7. Statements Regarding Scoring 1. I strongly disagree 3. I tend to disagree 5. I tend to agree 2. I disagree 4. I am undecided 6. I agree 7. I strongly agree. ) the score of the answers given to the question is added and divided by 9. If the result is less than 2.8, it is evaluated as "no fatigue". If the result is greater than 6.1, it is considered as "chronic fatigue syndrome
Pittsburgh Sleep Quality Index | 14 weeks
  It was developed by Buysse et al. (1989) (34). The scale is a safe and consistent questionnaire that evaluates the amount of sleep, sleep quality, presence and severity of sleep disorders in individuals in the last month. It was adapted into Turkish by Ağargün et al. (1996) (35). There are seven components in Pittsburg Sleep Quality Index. These components are subjective sleep quality (component 1), sleep latency (component 2), sleep duration (component 3), habitual sleep efficiency (component 4), sleep disturbance (component 5), sleep medication use (component 6) and daytime dysfunction. (component 7). The evaluation score of each item is between 0-3. The total score obtained varies between 0-21. The higher the score, the worse the sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Postacı, Study Chair — Uskudar University
Locations (1):
- Fizyorapt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozeren A, Ulug N, Sahan N, Can Karahan Z. Does reformer pilates exercise improve cognitive functions in sedentary women? A randomized controlled study. J Bodyw Mov Ther. 2024 Oct;40:1899-1905. doi: 10.1016/j.jbmt.2024.10.031. Epub 2024 Oct 18. PMID 39593541
- [Background] Aykut S, Sevgin O. Effect of video-based exercise on premenstrual symptoms: a randomized controlled trial. Ginekol Pol. 2025;96(2):102-108. doi: 10.5603/gpl.98199. Epub 2024 Oct 29. PMID 39469819
- [Background] Peinado AB, Alfaro-Magallanes VM, Romero-Parra N, Barba-Moreno L, Rael B, Maestre-Cascales C, Rojo-Tirado MA, Castro EA, Benito PJ, Ortega-Santos CP, Santiago E, Butragueno J, Garcia-de-Alcaraz A, Rojo JJ, Calderon FJ, Garcia-Bataller A, Cupeiro R. Methodological Approach of the Iron and Muscular Damage: Female Metabolism and Menstrual Cycle during Exercise Project (IronFEMME Study). Int J Environ Res Public Health. 2021 Jan 16;18(2):735. doi: 10.3390/ijerph18020735. PMID 33561085